CLINICAL TRIAL: NCT02204020
Title: Phase II Study of 5-azacytidine Maintenance After Allogeneic Hematopoietic Cell Transplantation for High-risk Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Brief Title: Phase II Study of 5-azacytidine Maintenance After Transplant for AML or MDS
Acronym: UPCI 13-165
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of interest with investigators - no subjects enrolled
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Annie Im, M.D., Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 13-165
Record Dates: First submitted 2014-07-25; First posted 2014-07-30 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS)
Keywords: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS); allogeneic; 5-azacytidine (5-aza); hematopoietic; transplantation; transplant; graft-versus-tumor; graft-versus-host disease (GVHD); epigenetic; maintenance; hypomethylation; relapse
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Graft vs Host Disease; Recurrence | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 5-azacytidine (Experimental): 5-aza SC or IV 32mg/m2 - 75mg/m2 (based on dose escalation)
  Interventions: Drug: 5-azacytidine (5-aza) maintenance therapy after transplant

INTERVENTIONS:
Drug: 5-azacytidine (5-aza) maintenance therapy after transplant — The planned initial dose of 5-aza is 32mg/m2 (Level 0) administered either subcutaneously or intravenously for days 1 through 5 of a 28-day cycle, which will be initiated between day+30 and day+100 after HCT. Patients who tolerate this dose based on hematologic parameters and with no SAEs for two consecutive cycles will be eligible for a dose escalation to 50mg/m2 (Level +1). Patients who tolerate this dose based on the same criteria as above for two consecutive cycles will be eligible for a dose escalation to 75mg/m² (Level +2). Patients will continue at dose Level +2 for the remainder of the study provided there are no toxicities that require dose reduction. Patients requiring a dose reduction are not eligible for re-escalation.
  Other Names: 5-aza

SUMMARY:
Despite improvements in outcomes after Hematopoietic Cell Transplantation (HCT) for Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS), the risk of relapse remains high and is the most common cause of mortality after HCT. Moreover, treatment options for relapse after HCT are limited. Strategies to reduce relapse with maintenance therapy in patients who are at high risk are needed to improve survival. 5-aza is a hypomethylating agent that has shown immune modulating properties that may enhance the graft-versus-leukemia (GVL) effect, including upregulation of tumor-associated antigen and costimulatory molecule expression. Moreover, 5-aza has properties that suggest protection against graft-versus-host disease (GVHD) as well. Preliminary data shows that it is well tolerated and effective in clinical use for the treatment of AML or MDS relapse after HCT, as well as for maintenance therapy. This study will evaluate the use of 5-aza for maintenance after HCT in patients with AML or MDS with risk factors that are associated with a high risk for relapse.

DETAILED DESCRIPTION:
Phase II study of 5-aza maintenance after allogeneic Hematopoietic Cell Transplantation (HCT) for high-risk Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS). Early studies indicate 5-aza is a hypomethylating agent that has shown immune modulating properties that may enhance the graft-versus-leukemia (GVL) effect, including upregulation of tumor-associated antigen and costimulatory molecule expression. 5-aza also has properties that suggest protection against graft-versus-host disease (GVHD). The primary objective is to evaluate relapse rate at one year. Secondary objectives will include the incidence of both acute and chronic GVHD as well as relapse-free survival, overall survival and toxicity. Correlatives will be performed to evaluate the effect of 5-aza maintenance on the immune system.

Subjects must be transplant candidates with MDS or high risk characteristics of AML. Subjects are consented, screened, then transplanted. Those showing complete response and no active GVHD after transplant can proceed to maintenance with 5-aza. Bone marrow biopsies are performed for response assessment after transplant as well as every three cycles (1 cycle=28 days) while on treatment. Dosing starts at 32mg/m2 and can be increased every 2 cycles without a serious adverse event (SAE), or reduced per toxicity for up to 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 with MDS or high-risk AML, morphologically confirmed and based on World Health Organization criteria (see below for definition of high-risk AML)*, who are transplant candidates with an available human leukocyte antigen (HLA) -matched sibling or unrelated donor with at least 8/8 match

  *Definition of high-risk AML:
* Age≥60 years
* Age<60 years with any of the following:

  * Secondary AML
  * Poor risk cytogenetics, which include abnormalities of chromosome 3, 5, or 7, trisomy 8, 11q23 abnormalities, t(6;9), 20q-, and complex karyotype
  * Fms-like tyrosine kinase 3 (FLT3) mutation
  * Disease status ≥ second complete remission (CR2) at time of HCT
  * Detectable disease at time of HCT
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate major organ function, as defined by AST and ALT < 2 x upper limit of normal, total serum bilirubin < 2 x upper limit of normal (unless due to hemolysis or Gilbert's syndrome, then no upper limit), creatinine < 2 x upper limit of normal, unless there is known chronic kidney disease (creatinine must be at baseline for subjects with chronic kidney disease)
* In agreement to use an effective barrier method of birth control to avoid pregnancy during the study and for a minimum of 30 days after study treatment, for all male and female patients who are fertile

Exclusion Criteria:

* Uncontrolled, life-threatening infection that is not responding to antimicrobial therapy
* Serum creatinine > 2 x upper limit of normal, unless there is known chronic kidney disease (creatinine must be at baseline for subjects with chronic kidney disease), aspartate aminotransferase (AST),alanine aminotransferase (ALT), or total bilirubin > 2x upper limit of normal
* History of psychiatric disorder which may compromise compliance with the protocol or which does not allow for appropriate informed consent
* Patient may not be receiving any other antineoplastic agents
* Pregnancy
* Concurrent use of any other investigational agents on a clinical trial
* Prior allogeneic stem cell transplant
* Known hypersensitivity to 5-azacytidine * Prior treatment with 5-azacytidine is allowed

Post-transplant eligibility and exclusion criteria

Patients will have to meet the following post-transplant eligibility criteria to initiate treatment:

* In complete response (including complete remission with incomplete blood count recovery and marrow complete response) on bone marrow biopsy for response assessment after HCT (typically day +30)
* Patient is within 30-100 days after HCT
* Absolute neutrophil count (ANC) ≥ 1000/µL, platelet count ≥ 20,000/µL
* ECOG performance status 0-2
* Adequate major organ function, as defined by AST and ALT < 2 x upper limit of normal, total serum bilirubin < 2 x upper limit of normal (unless due to hemolysis or Gilbert's syndrome, then no upper limit), creatinine < 2 x upper limit of normal unless there is known chronic kidney disease (creatinine must be at baseline for subjects with chronic kidney disease)
* In agreement to use an effective barrier method of birth control to avoid pregnancy during the study and for a minimum of 30 days after study treatment, for all male and female patients who are fertile

Patients may not have any of the following post-transplant exclusion criteria:

* Active grade II-IV acute GVHD, for example requiring treatment with steroids at a dose equivalent to prednisone 1mg/kg daily or higher
* Uncontrolled, life-threatening infection that is not responding to antimicrobial therapy
* Serum creatinine > 2 x upper limit of normal unless there is known chronic kidney disease (creatinine must be at baseline for subjects with chronic kidney disease), aspartate aminotransferase (AST),alanine aminotransferase (ALT), or total bilirubin > 2x upper limit of normal
* History of psychiatric disorder which may compromise compliance with the protocol or which does not allow for appropriate informed consent
* Pregnancy
* Concurrent use of any other investigational agents on a clinical trial
* Known hypersensitivity to 5-azacytidine * Prior treatment with 5-azacytidine is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2016-05-04 (Actual)

PRIMARY OUTCOMES:
Relapse rate at 1 year | 3 years
  Study will evaluate the relapse rate associated with 5-azacytidine (5-aza) as maintenance therapy after HCT in patients with high-risk AML or MDS.

SECONDARY OUTCOMES:
Safety of Toxicity Requiring Treatment Discontinuation (TRTD) | 3 years
Overall survival | 3 years
Incidence of acute GVHD | 3 years
Percentage of Toxicity Requiring Treatment Discontinuation (TRTD) | 3 years
relapse-free survival | 3 years
Incidence of chronic GVHD | 3 years

OTHER OUTCOMES:
Effect on the immune system | 3 years
  Study will evaluate the effect of 5-aza maintenance on the immune system using T-cell phenotype subsets and receptor expression, cytokine levels including tumor necrosis factor alpha (TNFα) and Interferon-y (IFNγ) (proinflammatory), and interleukin 7 (IL-7) and interleukin 15 (IL-15) (homeostatic) and association of correlative measures with relapse and incidence of GVHD.

CONTACTS AND LOCATIONS:
Overall Officials: Annie Im, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States